CLINICAL TRIAL: NCT04929496
Title: Physiology as Guidance to Evaluate the Direct Impact of Coronary Lesion Treatment: the PREDICT Study
Acronym: EASY-PREDICT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Opsens, Inc. (Industry); International Chair on Interventional Cardiology and Transradial Approach (Other)
Responsible Party: Principal Investigator, Olivier F. Bertrand, Study Principal Investigator, Laval University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: EASY-PREDICT pilot study
Record Dates: First submitted 2021-05-31; First posted 2021-06-18 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-01

CONDITIONS: Coronary Artery Disease; Stable Angina; Unstable Angina; Ischemic Heart Disease; Chest Pain
Keywords: Coronary Artery Disease; Fractional Flow Reserve; Post-PCI FFR; Angiography; Angioplasty
MeSH Terms: conditions — Coronary Artery Disease; Angina, Stable; Angina, Unstable; Myocardial Ischemia; Chest Pain | interventions — Fractional Flow Reserve, Myocardial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Angiographical guidance only (No Intervention): Standard of care
- Post-PCI FFR guidance (Experimental): Post-PCI Fractional Flow Reserve and non-hyperemic pressure ratios measurement
  Interventions: Procedure: post-PCI FFR

INTERVENTIONS:
Procedure: post-PCI FFR — final invasive physiology measurements after successful stent implantation, followed by functional optimization if physiology indexes remain positive.
  Other Names: Fractional Flow Reserve; Non-hyperemic pressure ratios
  Arms: Post-PCI FFR guidance

SUMMARY:
The purpose of this study is to assess whether the use of physiology parameters as guidance post-percutaneous coronary interventions (PCI) is associated with less risks of target vessel failure (TVF) and angina-related events than standard angiographic guidance.

DETAILED DESCRIPTION:
Fractional flow reserve (FFR) measurement involves determining the ratio between the maximum achievable blood flow in a diseased coronary artery and the theoretical maximal flow in a normal coronary artery. An FFR of 1.0 is widely accepted as normal. An FFR value less than or equal to 0.80 is generally considered to be associated with myocardial ischemia.

FFR is easily measured during routine coronary angiography by using a pressure wire to calculate the ratio between coronary pressure distal to a coronary artery stenosis and aortic pressure under conditions of maximum myocardial hyperemia. this ratio represents the potential decrease in coronary flow distal o the coronary stenosis. Recently, other physiology ratios called non-hyperemic ratios (NHPR) have been developed.

Both types of physiology measures (FFR and NHPR) have been increasingly used in cardiac catheterization laboratories as a diagnostic tool. They provide a quantitative assessment of the functional severity of a coronary artery stenosis identified during coronary angiography and cardiac catheterization. However, they are underutilized as tools for the assessment of success of coronary interventions.

The PREDICT study is a pilot study which aims to prospectively determine whether post-PCI physiology guidance is associated with better clinical outcomes than standard angiographic guidance.

ELIGIBILITY:
Inclusion Criteria:

* Any patient referred for diagnostic coronary angiography and / or possible PCI in native coronary vessels.
* Successful (< 30% diameter stenosis and normal TIMI 3 flow post-stenting) and uncomplicated PCI
* All treated lesions stented with drug-eluting stents (except side-branches of bifurcations)

Exclusion Criteria:

* Lesion in saphenous vein or arterial grafts
* Allergy to aspirin, thienopyridines or ticagrelor precluding treatment for 30 days
* Sub-optimal PCI result ( >30% residual diameter stenosis and/or <TIMI3 flow) or peri-procedural complications
* Acute ST-Elevation MI (culprit lesion)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Rate of Target Vessel Failure | within 18 months after index PCI;
  as the composite of cardiac death, lesion-related MI and target vessel revascularization
Rate of angina-related events | within 18 months after index PCI;
  defined as hospitalization for unstable angina and unsolicited medical visits for angina

SECONDARY OUTCOMES:
Final post-PCI pressure ratio values according to lesion location and intervened vessels | Post-randomization after stent implantation (< 1 hour)
  In the Physiology group, final pressure ratio (Pd/Pa) values will be collected immediately after randomization, and if further intervention is performed, before completing the intervention.
Final post-PCI FFR values according to lesion location and intervened vessels | Post-randomization after stent implantation (< 1 hour)
  In the Physiology group, final FFR values will be collected immediately after randomization, and if further intervention is performed, before completing the intervention.
Final post-PCI dPR values according to lesion location and intervened vessels | Post-randomization after stent implantation (< 1 hour)
  In the Physiology group, final dPR values will be collected immediately after randomization, and if further intervention is performed, before completing the intervention.
Final post-PCI physiology pullback curves according to lesion location and intervened vessels | Post-randomization after stent implantation (< 1 hour)
  In the Physiology group, final physiology pullback curves will be collected immediately after randomization, and if further intervention is performed, before completing the intervention if possible.
  Physiology pullback refers to either hyperemic or non-hyperemic pullback.
Rates of unstable angina requiring hospitalization or unsolicited medical visits | within 18 months of index procedure
Rates of individual components of MACE | within 18 months of index procedure
  including all-cause mortality, MI, TVR and any revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Olivier F. Bertrand, MD, PhD, Principal Investigator — International Chair on Interventional Cardiology and Transradial Approach
Locations (1):
- IUCPQ - Laval Hospital, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ulacia Flores P, Cieza T, Ouarrak S, Ruhl A, Mengi S, De Larochelliere R, Garcia-Labbe D, Dery JP, Poulin A, Larose E, Noel B, Nguyen CM, Paradis JM, Bertrand OF. Randomized Study Comparing Angiography Guidance With Physiology Guidance After PCI: The EASY-PREDICT Study. Circ Cardiovasc Interv. 2025 Jul;18(7):e015165. doi: 10.1161/CIRCINTERVENTIONS.125.015165. Epub 2025 May 21. PMID 40400236